CLINICAL TRIAL: NCT01834794
Title: Targeting Tobacco Cessation During Treatment for Cannabis Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Alan J. Budney, Professor, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 32243 D14201; 1R01DA032243-01 (NIH)
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Cannabis Dependence
Keywords: Tobacco Use
MeSH Terms: conditions — Marijuana Abuse; Tobacco Use | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MET/CBT/CM plus NRT (Experimental): Motivational Enhancement Therapy, Cognitive Behavior Therapy, Contingency Management plus Nicotine Replacement Therapy (MET/CBT/CM) + NRT
  Behavioral Treatment for Cannabis plus Behavioral Treatment for Tobacco: both primarily delivered by computer. Additional NRT.
  Interventions: Behavioral: MET/CBT/CM plus NRT

INTERVENTIONS:
Behavioral: MET/CBT/CM plus NRT — Behavioral Treatment for Cannabis plus Behavioral Treatment for Tobacco: both primarily delivered by computer. Additional NRT.

SUMMARY:
This project aims to develop and test an intervention for the simultaneous treatment of cannabis use disorders and tobacco smoking. This is important because over 50% of adults seeking treatment to help stop cannabis use also smoke tobacco regularly, which decreases their chance for a successful treatment outcome and increases adverse acute and long-term psychosocial and health consequences. The proposed treatment will integrate existing computer-based behavioral interventions for cannabis and tobacco and use nicotine replacement medications to improve outcomes in this difficult to treat clinical population.

DETAILED DESCRIPTION:
Approximately 50% of persons seeking treatment for cannabis-use disorders (CUDs) regularly smoke tobacco. Combining tobacco with cannabis has become a common method of smoking cannabis. Similarities of use, and using together, can make quitting difficult. Stopping tobacco simultaneously with cannabis may be beneficial. Little scientific information currently addresses how to best target tobacco smoking during treatment for CUDs. Our long-term goal is to develop an effective protocol for intervening in tobacco smoking without changing cannabis outcomes. A two-phase, Stage 1 therapy development project will accomplish the following: First, a treatment protocol and manual will be developed that integrates a tailored intervention for tobacco smoking with an intervention for CUD (Aim 1). Utilization of web-based counseling programs will standardize delivery of the intervention and foster eventual dissemination. A pilot study will provide an initial test of acceptability and feasibility. Second, a Stage 1, proof-of-concept study will compare this intervention to one that targets CUD only (Aim 2). The hypotheses assert that the intervention (1) will be accepted by the majority of eligible participants (2) will result in more tobacco quit attempts and rates than the CUD-only treatment; and (3) will not adversely affect cannabis outcomes. Last, the project will evaluate the potential of specific moderators of outcomes to predict outcomes and inform subsequent treatment development efforts (Aim 3). If the hypotheses were confirmed, dissemination of this protocol would reduce adverse psychosocial and health consequences of tobacco or cannabis dependence. Findings will inform future development of prevention and intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* current DSM-IV diagnosis of cannabis abuse or dependence
* report use of cannabis on at least 45 of previous 90 days
* report regular use of tobacco cigarettes or report that their primary administration of cannabis is via blunts or spliffs
* some indication of interest in quitting tobacco in the next 6 months (rating of 2 or more on a 5-point interest scale

Exclusion Criteria:

* current dependence on alcohol or any drug other than tobacco and cannabis
* active or recent suicidal ideation
* use of non-tobacco nicotine
* current participation in treatment for substance abuse
* severe psychological distress (e.g., active suicidal plans, psychosis, debilitating panic disorder).
* a condition that requires seeing a physician before using NRT (e.g., pregnancy or recent heart attack
* legal status that would interfere with participation
* living with someone enrolled in the project
* not living within 30 miles of the research site (unless an exception is authorized by the PI)
* not being fluent in english

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Tobacco Quit Attempts | Will be assessed for the duration of study, an average of 16 weeks
  Sum of 24 hour quit attempts

SECONDARY OUTCOMES:
Cannabis Abstinence: continuous weeks of abstinence achieved during the 12 week treatment period | Will be assessed twice per week for the duration of the study treatment period, 12 weeks
  Urinalysis tests and self-report data will be collected twice per week during participation in the study

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Budney, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - Geisel School of Medicine at Dartmouth; State Building Site, Concord, New Hampshire
  - Geisel School of Medicine at Dartmouth; Rivermill Complex Site, Lebanon, New Hampshire

REFERENCES:
- [Result] Lee DC, Budney AJ, Brunette MF, Hughes JR, Etter JF, Stanger C. Treatment models for targeting tobacco use during treatment for cannabis use disorder: case series. Addict Behav. 2014 Aug;39(8):1224-30. doi: 10.1016/j.addbeh.2014.04.010. Epub 2014 Apr 13. PMID 24813547